CLINICAL TRIAL: NCT06627062
Title: Intrascleral Fixation of Standard Capsular Tension Ring： a Modified-simple Technique for Managing Moderate and Severe Subluxated Lens Extraction
Brief Title: A Modified-simple Technique for Managing Moderate and Severe Subluxated Lens Extraction
Status: Completed | Type: Observational
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 202119
Record Dates: First submitted 2024-09-22; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Lens Subluxation
Keywords: Subluxated lens; Capsular bag; capsular tension ring; phacoemulsification
MeSH Terms: conditions — Lens Subluxation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- subluxated lens extraction: This research cohort consists of patients with moderate to severe subluxation who have successfully undergone lens extraction using an improved scleral fixation standard tension ring technique.
  Interventions: Procedure: moderate and severe subluxated lens extraction

INTERVENTIONS:
Procedure: moderate and severe subluxated lens extraction — A double-strand polypropylene suture (9-0 or 8-0) was looped and tied to one end of the preloaded CTR, which was then implanted into the capsular bag. The needle was inserted through the main incision, traversed the anterior chamber, under the posterior iris, and exited 2.0 mm behind the limbus at the central zonular weakness. The CTR was secured to the sclera using the knotless Z-suture technique to center the capsular bag, allowing safe insertion of the intraocular lens (IOL).
  Other Names: Intrascleral Fixation of Standard Capsular Tension Ring

SUMMARY:
The investigators describe a modified knotless Z-suture technique to stabilize the capsular bag to the sclera in eyes with moderate and severe ectopic lentis requiring cataract surgery using a standard CTR. This technology has the advantages of few complications, low technical difficulty, and no dependence on complex equipment.

DETAILED DESCRIPTION:
A dislocated crystalline lens, also known as ectopia lentis, is the result of lax zonule fibers causing the lens to dislocate from its anatomical position, which can be caused by various factors such as inherited autosomal dominant disorders, trauma, or several systemic diseases. According to the ratio of the pupil area uncovered by the lens to the whole pupil area after mydriasis, the degree of subluxation of the crystalline lens can be divided into three grades: mild (0-25%), moderate (25-50%), and severe (more than 50%). Moderate or severe cases may manifest as progressive blurred vision, monodiplopia or even secondary angle-closure glaucoma, resulting in a poor prognosis, thereby emphasizing the urgency for effective therapeutic interventions. Preserving the posterior capsular diaphragm is the key to preventing glaucoma, optic capture, and retinal detachment.

Phacoemulsification and fixation of the capsular bag have been described with various methods and devices, such as intraoperative use of iris hooks orcapsular retractors, and permanent capsular support like Capsular tension rings (CTRs) firstly introduced in 1993 by Legler et al6. It is recommended to use a standard CTR when the zonular weakness is less than 120 degrees (<4 clock hours). However, in instances of more extensive zonular weakness and progressive pathologies such as Marfan syndrome, Weill-Marchesani syndrome, pseudo exfoliation, high myopia and homocystinuria, intrascleral fixation of the capsular bag with a capsular tension segment (CTS), a modified CTR (m-CTR) or other devices such as the Assia Anchor is recommended6. However, m-CTR and a variety of new capsule assist devices are difficult to obtain in some countries. Therefore, how to make the most of the common auxiliary tools such as standard CTR in moderate and severe subluxation to retain the capsular bag requires ophthalmologists to continue exploring.

The investigators describe a novel technique of stabilizing a moderate or severe subluxated capsular bag which utilizes double-strand polypropylene sutures to suspend a standard capsular tension ring thereby enabling safe insertion of an intraocular lens (IOL) within the bag. The technique has been successfully demonstrated in 16 eyes of nine patients with congenital or traumatic lens subluxations ranging between 120 and 300 degrees.

ELIGIBILITY:
Inclusion Criteria:

- Patients with moderate to severe lens subluxation ranging from 120-300 degrees caused by different reasons.

Exclusion Criteria:

- Unable to cooperate in completing the lens subluxation surgery Lens subluxation accompanied by eyeball rupture injury Refuse surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The technique was successfully used in 16 eyes of 9 patients (including 3 females and 6males) with 15 congenital and 1 traumatic lens subluxations with subluxation ranges between 120-300 degrees.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Success rate of intraocular lens implantation in patients with moderate to severe subluxation of the crystalline lens | From enrollment to the end of treatment at 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Yinghong Ji, Phd; MD, Principal Investigator — Eye & ENT Hospital, Fudan University
Locations (1):
- Eye Institute and Department of Ophthalmology, Eye & ENT Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ning L, Hong Y, Ji Y. Intrascleral fixation of standard capsular tension ring: a modified-simple technique for managing moderate and severe subluxated lens extraction. Ther Adv Ophthalmol. 2026 Jan 27;18:25158414251407874. doi: 10.1177/25158414251407874. eCollection 2026 Jan-Dec. PMID 41613822